CLINICAL TRIAL: NCT00807378
Title: Cerebrospinal Fluid Polymerase Chain Reaction Arrays for Central Nervous System Neurotropic Viral Infection and Mycobacterium Infection Study
Brief Title: Rijavithi Viral and Mycobacterium PCR Arrays in CNS Infection Study
Acronym: VIMPAC
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Rajavithi Biomolecular Research Center (Other)
Responsible Party: Piyathida Harnsomboonrana, Rajavithi Biomolecular Research Center
Other Study IDs: RH-CMR-004
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: CNS Viral Infection
Keywords: CNS viral infection; PCR; HYBRIDIZATION
MeSH Terms: conditions — Central Nervous System Viral Diseases | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CSF DNA/RNA virus
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: AIDS PATIENTS
  Interventions: Other: LUMBAR PUNCTURE
- 2: NON-AIDS PATIENTS
  Interventions: Other: LUMBAR PUNCTURE

INTERVENTIONS:
Other: LUMBAR PUNCTURE — LUMBAR PUNCTURE FFOR CSF COLLECTION

SUMMARY:
This study of neurotropic viral infection and Tuberculous CNS infection is the comprehensive investigation of CSF PCR arrays (Hybrydiaztion technique,Sybergreen and Taqman real time PCR arrays of CSF ) in suspected cases of viral CNS infection, Tuberculous CNS infection in both AIDS and non AIDS patients.

Patients with clinical viral encephalitis and all meningoencephalitis including all patients with HIV/AIDS CSF and non AIDS will be banked and test for RNA and DNA viral sequence by Real time PCR arrays and IS6110 gene of Mycobacterium tuberculosis. Clinical data and final diagnosis will be used to analyze the result of this PCR arrays technique compared to clinical gold standard criteria.

ELIGIBILITY:
Inclusion Criteria:

1. AGE MORE THAN 15 YRS
2. ABLE TO INFORM CONSENT BY THEMSELF OR THEIR PARENT
3. SUSPECTED CNS VIRAL INFECTION

Exclusion Criteria:

1. UNABLE/CONTRAINDICATED FOR LUMBAR PUNCTURE OR CSF COLLECTION
2. WITHDRAW CONSENT
3. SUSPECTED SEVERE OR VILURENT VIRAL INFECTION SUCH AS H5N1/SARS INFECTION

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CNS VIRAL INFECTION AIDS/NON-AIDS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)